CLINICAL TRIAL: NCT01163279
Title: Maintaining Autonomy as we Age: Investigating the Application of a Strategy Training Approach for Ameliorating the Effects of Age-related Executive Dysfunction - Part II
Brief Title: Maintaining Autonomy as we Age. Strategy Training for Age-related Executive Dysfunction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baycrest (Other)
Responsible Party: Principal Investigator, Dr. Deirdre Dawson, Senior Scientist, Baycrest
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: REB1021
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Results first posted 2017-01-12 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-11

CONDITIONS: Aging
Keywords: Age-related changes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Training (Experimental)
  Interventions: Behavioral: Real world strategy approach
- Psychosocial Education (Active Comparator)
  Interventions: Behavioral: Psychosocial Education

INTERVENTIONS:
Behavioral: Real world strategy approach — The key features of the protocol are: i. Participants are actively engaged in selecting their treatment goals. The research clinician will work with the participants to identify five specific, measurable real-world goals using a standardized semi-structured interview, the Canadian Occupational Performance Measure. Three of these will be training goals, two will not be trained but evaluated post-intervention for evidence of generalization and transfer to non-trained tasks; ii. A global problem solving approach is used (Goal- Plan- Do- Check). Participants are guided by the trainer to apply this strategy to their goals.
  Other Names: Adopted Cognitive Orientation to Occupational Performance (CO-OP)
  Arms: Cognitive Training
Behavioral: Psychosocial Education — The active comparator uses an information-based format and is designed to engage participants without providing any specific training techniques or strategies. During weekly sessions, participants will receive factual information on brain structure and function, age-related cognitive changes, and general brain health issues and will spend time doing non-specific cognitive exercises including crossword and Sudoku puzzles. Homework will consist of reading assignments related to the session topics.
  Arms: Psychosocial Education

SUMMARY:
Healthy older adults with self-reported cognitive difficulties who receive strategy training will demonstrate greater performance benefits on measures of real-world activities, relative to those receiving a control intervention, immediately post treatment and at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All participants must score within 1.5 standard deviation (SD) of age and education-corrected normative data for the Montreal Cognitive Assessment and on a battery of neuropsychological tests of attention, memory and executive function (which will insure that participants are unlikely to meet the criteria for Mild Cognitive Impairment (MCI)).
* No clinically relevant depression (scores ≤22) on the Center for Epidemiologic Studies Depression Scale (CES-D)
* Fluent in written and spoken English
* Self-reported complains about cognitive function

Exclusion Criteria:

* Recent bereavement (within last 6 months)
* History of neurological disease
* Psychiatric illness requiring hospitalization and/or history or current substance abuse

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Dawson, PhD, Principal Investigator — Rotman Research Institute, Baycrest
Locations (1):
- Baycrest, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a research subject pool and a community psycho-education program at Baycrest.
Pre-assignment Details: A total of 96 participants were assessed for study eligibility. 60 participants were excluded after a phone screening interview and 17 were excluded after a more detailed baseline assessment which included cognitive paper and pencil tasks. The remaining 19 participants were randomized to either the experimental arm or the control arm.
Groups:
- Cogntive Training: Real world strategy approach: The key features of the protocol are: i. Participants are actively engaged in selecting their treatment goals. The research clinician will work with the participants to identify five specific, measurable real-world goals using a standardized semi-structured interview, the Canadian Occupational Performance Measure. Three of these will be training goals, two will not be trained but evaluated post-intervention for evidence of generalization and transfer to non-trained tasks; ii. A global problem solving approach is used (Goal- Plan- Do- Check). Participants are guided by the trainer to apply this strategy to their goals.
- Psychosocial Education: The active comparator was an information-based format and is designed to engage participants without providing any specific training techniques or strategies. During weekly sessions, participants received factual information on brain structure and function, age-related cognitive changes, and general brain health issues and spent time doing non-specific cognitive exercises including crossword and Sudoku puzzles. Homework consisted of reading assignments related to the session topics.
Period: Overall Study
Arm/Group | Cogntive Training | Psychosocial Education
Started | 10 | 9
Completed | 8 | 9
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Training | Psychosocial Education | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.10 (8.77) | 73.67 (5.43) | 73.94 (7.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Goals Improved to Criterion on the Canadian Occupational Performance Measure (COPM)
Description: COPM is a standardized semi-structure interview in which participants identify goals related to everyday life activities. Goals considered improved to criterion are those that had 2 or more points increase on COPM ratings.
Time Frame: Immediately post intervention (2 months) and 3 months later
Population: Intention to treat analysis was done therefore, the analysis population includes all participants who were randomized (n=19).
Measure: Number; unit: percentage of untrained goals improved
Units Other Than Participants: Total number of goals
Arm/Group | Cognitive Training | Psychosocial Education
Number analyzed (Participants) | 10 | 9
Number analyzed (Total number of goals) | 52 | 46
percentage of untrained goals improved
  post intervention performance | 50 | 19.6
  post intervention satisfaction | 50 | 32.6
  3-month follow up performance | 36.4 | 26.1
  3-month follow up satisfaction | 45.5 | 28.3
Statistical Analysis 1: Comparison: Cognitive Training vs Psychosocial Education; Test type: Superiority or Other; p = 0.03, Chi-squared — Statistical analysis applies to post intervention performance category
Statistical Analysis 2: Comparison: Cognitive Training vs Psychosocial Education; Test type: Superiority or Other; p = 0.32, Chi-squared — Statistical analysis applies to post intervention satisfaction category
Statistical Analysis 3: Comparison: Cognitive Training vs Psychosocial Education; Test type: Superiority or Other; p = 0.54, Chi-squared — Statistical analysis applies to 3-month follow up performance category
Statistical Analysis 4: Comparison: Cognitive Training vs Psychosocial Education; Test type: Superiority or Other; p = 0.26, Chi-squared — Statistical analysis applies to 3-month follow up satisfaction category

2. Secondary Outcome: General Self Efficacy Scale (GSE)
Description: GSE is a self efficacy scale with a minimum score of 10 and a maximum score of 40. Higher scores indicate higher self efficacy
Time Frame: Baseline, Immediately post intervention (2 months) and 3 months later
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Cognitive Training | Psychosocial Education
Number analyzed (Participants) | 10 | 9
Scores on scale
  Baseline | 29.10 (3.41) | 32.56 (3.40)
  Immediately post intervention (2 months) | 30.90 (3.98) | 33.56 (4.28)
  3 months post intervention | 30.50 (4.12) | 33.56 (3.43)
Statistical Analysis 1: Comparison: Cognitive Training vs Psychosocial Education; Test type: Superiority or Other; p < 0.05, ANOVA — Statistical analysis applies to immediately post intervention and 3 months post intervention categories

3. Secondary Outcome: Stanford Patient Education Research Center- General Health Subscale
Description: Stanford Patient Education Research Center has different measures of health related behaviors. General Health is one of the subscales. scores range 1-5 and higher score indicate better general health
Time Frame: Baseline, Immediately post intervention (2 months) and 3 months later
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training | Psychosocial Education
Number analyzed (Participants) | 10 | 9
units on a scale
  Baseline | 2.20 (0.63) | 1.89 (0.78)
  Immediately post intervention (2 months) | 2.20 (0.42) | 1.78 (0.83)
  3 months post intervention | 2.20 (0.92) | 2.00 (0.87)
Statistical Analysis 1: Comparison: Cognitive Training vs Psychosocial Education; Test type: Superiority or Other; p > 0.05, ANOVA — Statistical analysis applies to immediately post intervention and 3 months post intervention categories

4. Secondary Outcome: Stanford Patient Education Research Center- Health Distress Subscale
Description: Stanford Patient Education Research Center has different measures of health related behaviors. Health distress is one of the subscales. Scores range 0-20 and higher score indicates more distress.
Time Frame: Baseline, Immediately post intervention (2 months) and 3 months later
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training | Psychosocial Education
Number analyzed (Participants) | 10 | 9
units on a scale
  Baseline | 2.70 (2.21) | 4.22 (2.77)
  Immediately post intervention (2 months) | 3.80 (3.46) | 3.67 (4.21)
  3 months post intervention | 3.70 (3.37) | 4.11 (2.03)
Statistical Analysis 1: Comparison: Cognitive Training vs Psychosocial Education; Test type: Superiority or Other; p > 0.05, ANOVA — Statistical analysis applies to immediately post intervention and 3 months post intervention categories

5. Secondary Outcome: Stanford Patient Education Research Center- Physical Activity Subscale
Description: Stanford Patient Education Research Center has different measures of health related behaviors. Physical activity is one of the subscales. Scores indicate number of hours of physical activity per week
Time Frame: Baseline, Immediately post intervention (2 months) and 3 months later
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours of physical activity/week
Arm/Group | Cognitive Training | Psychosocial Education
Number analyzed (Participants) | 10 | 9
hours of physical activity/week
  Baseline | 4.08 (2.22) | 5.31 (1.47)
  Immediately post intervention (2 months) | 4.45 (2.53) | 3.64 (1.35)
  3 months post intervention | 4.15 (1.83) | 3.19 (1.56)
Statistical Analysis 1: Comparison: Cognitive Training vs Psychosocial Education; Test type: Superiority or Other; p < 0.05, ANOVA — Statistical analysis applies to immediately post intervention and 3 months post intervention categories

6. Secondary Outcome: Stanford Patient Education Research Center- Communication With Physicians Subscale
Description: Stanford Patient Education Research Center has different measures of health related behaviors. communication with physicians is one of the subscales. Scores range 1-15 and higher score indicates more preparation for visits and greater ability to ask questions
Time Frame: Baseline, Immediately post intervention (2 months) and 3 months later
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training | Psychosocial Education
Number analyzed (Participants) | 10 | 9
units on a scale
  Baseline | 8.40 (3.84) | 11.00 (3.04)
  Immediately post intervention (2 months) | 9.50 (4.17) | 9.11 (3.33)
  3 months post intervention | 10.00 (3.80) | 8.89 (4.17)
Statistical Analysis 1: Comparison: Cognitive Training vs Psychosocial Education; Test type: Superiority or Other; p < 0.1, ANOVA — Statistical analysis applies to immediately post intervention category
Statistical Analysis 2: Comparison: Cognitive Training vs Psychosocial Education; Test type: Superiority or Other; p < 0.05, ANOVA — Statistical analysis applies to 3 months post intervention category

7. Secondary Outcome: Stanford Patient Education Research Center- Visits to Physician and Emergency Department in the Past Six Months Subscale
Description: Stanford Patient Education Research Center has different measures of health related behaviors. Visits to physician and emergency department in the past six months subscale is one of the subscales.
Time Frame: Baseline, Immediately post intervention (2 months) and 3 months later
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Cognitive Training | Psychosocial Education
Number analyzed (Participants) | 10 | 9
number of visits
  Baseline | 2.30 (0.95) | 2.78 (3.07)
  Immediately post intervention (2 months) | 1.50 (0.97) | 3.33 (4.00)
  3 months post intervention | 2.00 (1.24) | 2.33 (2.74)
Statistical Analysis 1: Comparison: Cognitive Training vs Psychosocial Education; Test type: Superiority or Other; p < 0.05, ANOVA — Statistical analysis applies to immediately post intervention category
Statistical Analysis 2: Comparison: Cognitive Training vs Psychosocial Education; Test type: Superiority or Other; p > 0.05, ANOVA — Statistical analysis applies to 3 months post intervention category

8. Secondary Outcome: Delis Kaplan Executive Function System (DKEFS) Tower Test- Mean First-Move Time
Description: This is a measure of executive function. The score reflects the average of the participant's first-move times, i.e. the time a participant took to make the first move
Time Frame: Baseline, Immediately post intervention (2 months) and 3 months later
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Time in seconds
Arm/Group | Cognitive Training | Psychosocial Education
Number analyzed (Participants) | 10 | 9
Time in seconds
  Baseline | 5.48 (3.72) | 6.13 (5.83)
  Immediately post intervention (2 months) | 3.00 (1.72) | 3.69 (2.89)
  3 months post intervention | 2.47 (1.78) | 1.72 (0.71)
Statistical Analysis 1: Comparison: Cognitive Training vs Psychosocial Education; Test type: Superiority or Other; p < 0.1, ANOVA — Statistical analysis applies to immediately post intervention category
Statistical Analysis 2: Comparison: Cognitive Training vs Psychosocial Education; Test type: Superiority or Other; p < 0.05, ANOVA — Statistical analysis applies to 3 months post intervention category

9. Secondary Outcome: DKEFS Tower Test- Achievement Score
Description: This is a measure of executive function. Total achievement scores indicate the highest score participants scored on the test. The lowest score possible is 0 and the highest score possible is 30. Higher scores indicate better performance.
Time Frame: Baseline, Immediately post intervention (2 months) and 3 months later
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training | Psychosocial Education
Number analyzed (Participants) | 10 | 9
units on a scale
  Baseline | 17.10 (3.57) | 15.78 (4.09)
  Immediately post intervention (2 months) | 18.30 (3.59) | 19.44 (4.07)
  3 months post intervention | 20.90 (4.31) | 18.89 (3.30)
Statistical Analysis 1: Comparison: Cognitive Training vs Psychosocial Education; Test type: Superiority or Other; p < 0.05, ANOVA — Statistical analysis applies to immediately post intervention and 3 months post intervention categories

10. Secondary Outcome: DKEFS Word Fluency
Description: This is a measure of executive function where participants are given a letter and asked to generate as many words as they can think of within 60 seconds
Time Frame: Baseline, Immediately post intervention (2 months) and 3 months later
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of words generated
Arm/Group | Cognitive Training | Psychosocial Education
Number analyzed (Participants) | 10 | 9
Number of words generated
  Baseline | 55.30 (15.25) | 48.56 (11.74)
  Immediately post intervention (2 months) | 56.40 (18.38) | 50.33 (9.12)
  3 months post intervention | 57.40 (16.34) | 50.11 (13.05)
Statistical Analysis 1: Comparison: Cognitive Training vs Psychosocial Education; Test type: Superiority or Other; p > 0.05, ANOVA — Statistical analysis applies to immediately post intervention category
Statistical Analysis 2: Comparison: Cognitive Training vs Psychosocial Education; Test type: Superiority or Other; p < 0.05, ANOVA — Statistical analysis applies to 3 months post intervention category

11. Secondary Outcome: DKEFS Trail Making- Condition 4: Number-letter Switching
Description: DKEFS trail making condition 4 is a measure of executive function that requires the participant to switch back and forth between connecting numbers and letters in a sequence
Time Frame: Baseline, Immediately post intervention (2 months) and 3 months later
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Time in seconds
Arm/Group | Cognitive Training | Psychosocial Education
Number analyzed (Participants) | 10 | 9
Time in seconds
  Baseline | 104.50 (43.87) | 91.11 (19.19)
  Immediately post intervention (2 months) | 88.40 (28.55) | 80.56 (25.37)
  3 months post intervention | 94.10 (32.70) | 84.44 (31.33)
Statistical Analysis 1: Comparison: Cognitive Training vs Psychosocial Education; Test type: Superiority or Other; p > 0.05, ANOVA — Statistical analysis applies to immediately post intervention and 3 months post intervention categories

ADVERSE EVENTS:
Time Frame: 2 months-during the intervention phase of the study
Groups:
- Psychosocial Education: Real world strategy approach: The key features of the protocol are: i. Participants are actively engaged in selecting their treatment goals. The research clinician will work with the participants to identify five specific, measurable real-world goals using a standardized semi-structured interview, the Canadian Occupational Performance Measure. Three of these will be training goals, two will not be trained but evaluated post-intervention for evidence of generalization and transfer to non-trained tasks; ii. A global problem solving approach is used (Goal- Plan- Do- Check). Participants are guided by the trainer to apply this strategy to their goals.
Arm/Group | Cognitive Training | Psychosocial Education
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No